CLINICAL TRIAL: NCT06234189
Title: The Immediate Effect of Defocus Incorporated Multiple Segment Spectacle Lenses (DIMS) on the Choroid Thickness Using Swept Source-Optical Coherence Tomography (SS-OCT) on Children.
Brief Title: The Immediate Effect of Defocus Spectacles On the Choroid Thickness Using Optical Coherence Tomography on Children
Acronym: TIDOCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TIDOCT
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Defocus Incorporated Multiple Segment Spectacle Lenses (DIMS) (Experimental)
  Interventions: Device: Defocus Incorporated Multiple Segment Spectacle Lenses (DIMS)

INTERVENTIONS:
Device: Defocus Incorporated Multiple Segment Spectacle Lenses (DIMS) — 30 minutes without DIMS and 30 minutes with DIMS

SUMMARY:
The purpose is to examine temporary changes in the subfoveal choroid thickness after removal and after resumed use of Defocus Incorporated Multiple Segment Spectacle Lenses (DIMS).

ELIGIBILITY:
Inclusion Criteria:

* Myopic children using Defocus Incorporated Multiple Segment Spectacle Lenses (DIMS) from the ongoing randomized clinical non-inferiority study: "Defocus Incorporated Multiple Segment (DIMS) Spectacle Lenses versus Orthokeratology lenses (OKL) for slowing myopia progression in children aged 6-12 years. A non-inferiority randomized clinical trial. The NISDO study" (ClinicalTrials.gov Identifier NCT05134935).
* Myopia at the time of inclusion in the NISDO study (inclusive): -2.00 to -4.75 D spherical component and up to -2.50 D of regular astigmatism (both eyes).
* Anisometropia at the time of inclusion in the NISDO study ≤ 1.50 D cycloplegic spherical equivalent refractive error.
* Best corrected visual acuity (inclusive) at the time of inclusion in the NISDO study: 0.8 Snellen (equivalent to ≥ 3/5 letter on the 0.8 line = 78 ETDRS letters).

Exclusion Criteria:

* Manifest or intermittent squint.
* Contraindications to the use of OKL comprising (not exhaustive): keratoconus, chronic allergic conjunctivitis, and keratoconjunctivitis sicca.
* Previous eye surgery.
* Chronic eye disease demanding daily use of eye drops.
* Non-compliance to eye examinations (unstable fixation or anxiety towards contact lenses).
* Previous myopia control treatment.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | During 60 minutes
  Thickness is measured in um

CONTACTS AND LOCATIONS:
Overall Officials: Lou-Ann Andersen, Principal Investigator — Vejle Hospital
Locations (1):
- The Ophthalmic department, Vejle Hospital, Vejle, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT06234189/SAP_001.pdf